CLINICAL TRIAL: NCT05674318
Title: Evaluation of Prebiotic Effects of Alpha-lactalbumin on Microbiota Composition
Brief Title: The Effect of Alpha-lactalbumin on Microbiota Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PREBIO_LAC22
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-06

CONDITIONS: Alpha-lactalbumin; Microbiota; Dysbiosis
MeSH Terms: conditions — Dysbiosis | interventions — Lactalbumin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpha-lactalbumin (Experimental)
  Interventions: Dietary Supplement: Alpha-lactalbumin

INTERVENTIONS:
Dietary Supplement: Alpha-lactalbumin — Oral assumption of two tabs/day containing Alpha-lactalbumin for 30 days

SUMMARY:
To evaluate the effects on microbiota composition after the administration of an oral supplementation based on Alpha-lactalbumin in subjects with dysbiosis.

ELIGIBILITY:
Inclusion Criteria:

* condition of dysbiosis

Exclusion Criteria:

* antibiotic treatment within 1 month
* probiotic or prebiotic treatments
* concomitant inflammatory intestinal diseases
* pregnancy
* neoplastic diseases
* allergy to milk protein (Alpha-lactalbumin)
* substance abuse

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement of microbiota composition | Change from baseline microbiota composition to 30 days of treatment
  Determination of bacterial biodiversity by metagenomics approach

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Polispecialistico Giovanni Paolo I°, Viterbo, Rome, Italy